CLINICAL TRIAL: NCT00269165
Title: Adjuvant Radiation in Aortic Valvuloplasty - ARAVA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005-187
Record Dates: First submitted 2005-12-22; First posted 2005-12-23 (Estimated); Last update posted 2010-05-31 (Estimated); Status verified 2010-05

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

INTERVENTIONS:
Procedure: Balloon Aortic Valvuloplasty
Procedure: External Beam Radiation

SUMMARY:
This study will examine the effect of external beam radiation therapy in the prevention of restenosis following successful balloon aortic valvuloplasty in severe, symptomatic aortic stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Severe Aortic Stenosis
* NYHA Class 2-4 CHF Symptoms
* Age > 75
* EuroSCORE > 7
* Prohibitively High Risk for Aortic Valve Replacement Surgery as Designated by a Cardiac Surgeon

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60
Dates: Start 2005-11

CONTACTS AND LOCATIONS:
Overall Officials: Ron Waksman, MD, Principal Investigator — Medstar Health Research Institute